CLINICAL TRIAL: NCT02974478
Title: Impact of Orange Juice Consumption on Glucose Homeostasis and Antioxidative Status in Healthy Subjects
Brief Title: Orange Juice Consumption and Glucose Metabolism and Antioxidative Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OrangeJuice
Record Dates: First submitted 2016-11-02; First posted 2016-11-28 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: orange juice consumption; glucose homeostasis; antioxidative status
MeSH Terms: interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Orange juice with meals (Experimental): Effect of orange juice consumption with three meals per day (without snacking) on glucose metabolism and antioxidative status
  Interventions: Dietary Supplement: Orange juice with meals
- Orange juice between meals (Experimental): Effect of orange juice consumption between three meals per day (without snacking) on glucose metabolism and antioxidative status
  Interventions: Dietary Supplement: Orange juice between meals
- Sugar sweetened beverage between meals (Experimental): Effect of sugar sweetened beverage consumption between three meals per day (without snacking) on glucose metabolism and antioxidative status
  Interventions: Dietary Supplement: Sugar sweetened beverage between meals

INTERVENTIONS:
Dietary Supplement: Orange juice with meals — orange juice (20% of energy requirement/day)
  Arms: Orange juice with meals
Dietary Supplement: Orange juice between meals — orange juice (20% of energy requirement/day)
  Arms: Orange juice between meals
Dietary Supplement: Sugar sweetened beverage between meals — Sugar sweetened beverage (20% of energy requirement/day)
  Arms: Sugar sweetened beverage between meals

SUMMARY:
Aim of the study is to investigate the impact of orange juice consumption (with meals or between meals) as well as sugar sweetened beverage (SSB) consumption (between meals) on glucose homeostasis and antioxidative status.

DETAILED DESCRIPTION:
Duration of the study is 3x three weeks including one wash-out week each followed by two weeks of juice/SSB consumption under free living conditions.

During wash-out weeks consumption of orange juice or citrus fruits is restricted.

During intervention weeks, participants are asked to eat three regular meals per day without snacking. Intervention weeks are (i) orange juice consumption with meals (ii) orange juice consumption between meals and (iii) SSB consumption between meals. Daily energy intake with orange juice/SSB is 20% of individual energy requirement. Additional caloric beverages (SSB, juice, coffee with sugar/milk, alcohol) are not allowed. At the beginning and the end of each intervention phase insulin sensitivity and antioxidative status are assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* regular use of medication,
* smoking,
* chronic disease,
* vegan/vegetarian diet,
* fructose intolerance,
* irregular eating behaviour (less then 3 meals/day)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
changes in daylong glycaemia between pre and post intervention periods | two weeks
  measured via continuous glucose monitoring [mg/dL]

SECONDARY OUTCOMES:
changes in uric acid between pre and post intervention periods | two weeks
  measured via uric acid serum levels [mg/dL]
changes in insulin sensitivity between pre and post intervention periods | two weeks
  measured via "Matsuda-Index" from oral glucose tolerance test data
changes in antioxidative status between pre and post intervention periods | two weeks
  measured via vitamin c blood levels [mg/L]

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, Prof PhD, Principal Investigator — University of Hohenheim, Stuttgart, Germany
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No